CLINICAL TRIAL: NCT01419522
Title: Effect of Time Varying Walking Velocity in Body-Weight Supported Treadmill Training
Brief Title: Treadmill Training at Constant or Different Speeds for People With Traumatic Brain Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 110203; 11-CC-0203
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-01-06

CONDITIONS: Traumatic Brain Injury; Walking Impairment; Gait Training
Keywords: Traumatic Brain Injury; Walking Impairment; Gait Training; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

INTERVENTIONS:
Other: Gait Training Method — Treadmill training at constant velocity

SUMMARY:
Background:

- Many people who have had a traumatic brain injury have difficulty walking. Training on a treadmill is often used to help people with walking difficulties. Supporting a person s body weight with a harness while using the treadmill can help improve walking skills in people with brain injury. Varying the rate at which people walk on the treadmill may also help more than walking at a constant rate. Treadmill training with body weight support or walking at different speeds may improve walking skills in people who have had a traumatic brain injury. More research is needed to see if one method is better than the other.

Objectives:

- To compare the effects of two types of treadmill training in people who have had a traumatic brain injury.

Eligibility:

- People at least 18 years of age who have had a mild or moderate traumatic brain injury at least 6 months ago and have mild or moderate walking difficulty.

Design:

* Participants will be screened with a medical history and physical exam. They will also take a basic walking test (not on a treadmill).
* Participants will be divided into two groups. The first group will have treadmill training at a constant speed. The second group will have treadmill training at different speeds. All participants will wear a support harness while walking on the treadmill.
* At the first training visit, participants will have a gait assessment with different tests of walking. Then they will have a treadmill walking session.
* After the first visit, participants will return twice a week for 6 weeks for treadmill training sessions (visits 3 through 12). They will also have grip strength and walking tests.
* At the end of 6 weeks, participants will have a final treadmill training session, and will have a gait assessment exactly like the one in the first training visit.
* At 6 months after the final session, participants will have a followup visit with a final gait assessment.

DETAILED DESCRIPTION:
Objectives: To test the effectiveness of using time varying walking velocity in Body-Weight Supported Treadmill Training (BWSTT) as compared to using constant velocity in subjects with Traumatic Brain Injury (TBI). We hypothesize that using time varying velocity will result in a greater improvement in ambulatory function.

Study Population: 30 adult subjects with a clinical diagnosis of non-penetrating TBI and with functional deficits in gait will be enrolled. Subjects will be recruited from NIH, affiliated hospitals/clinics, and in the community.

Design: This pilot study will use an instrumented treadmill (Bertec Co., Columbus, Ohio) and a force controlled harness system called ZeroG (Aretech LLC, Ashburn, Virginia). Subjects will be randomly assigned to one of two groups (12 subjects per group): the first group will receive BWSTT at a constant velocity (also known as standard treadmill training); and the second group will receive BWSTT at randomized time varying velocity. BWSTT at time varying velocity consists of two components: 1) subjects passively adjusting their walking speed to the continuously changing speed of the treadmill; and 2) subjects actively changing their walking speed by following the instructed walking speed displayed on a monitor screen while the treadmill is automatically adjusted to the subjects speed. Each group will receive 8 gait training sessions (30 minutes per session, twice per week) for four weeks. Gait performance will be tested before (pre-test) and after (post-test) the 8 session gait training program.

Outcome Measures: The primary outcome measures are parameters representing gait performance: maximum walking speed, self-selected walking speed, cadence, stride length, percentage of swing, stance and double stance periods, gait symmetry, Time Up and Go (TUG), and Dynamic Gait Index (DGI) scores. The secondary outcome measure is physical and cognitive effort exerted during the training session as evaluated by grip-strength test and LNS (Letter-Number Sequencing) test.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects eligible for participation in this research study must meet the following inclusion criteria:

Diagnosis of non-penetrating TBI, specifically functionally mild to moderate TBI (those individuals who demonstrate the ability or capacity to ambulate)

Injury occurred at least 6 months prior to enrollment

Age of 18 or older

Able to stand and walk on a treadmill for 30 minutes (with some breaks in the middle)

Have mild or moderate functional gait impairment (score 1 or 2 in the first two tests in DGI: 1. Gait Level Surface test and 2. Change in Gait Speed test)

Able to provide informed consent

Able to read 3 inch by 3 inch letters in the monitor located at 1 meter distance from the treadmill without affecting gait patterns on the treadmill.

EXCLUSION CRITERIA:

Subjects are not eligible for participation in this research study if any of the following conditions exist:

Taking medications that affect motor function such as baclofen, levodopa, benzodiazepams, tizanadine, or dantrolene sodium.

Had surgery to either lower limb within the last year or requires surgery during the period of the study

Had botulinum toxin injections in lower limbs within the last 4 months or willing to forego botulinum toxins in lower limbs for the duration of the study

Are currently receiving any type of gait training or similar intervention outside of the study or unwilling to forego initiation of such an intervention during the period of this study

Presence of severe pain in the lower limbs (VAS 5 or above)

Medical or psychological instability such that the clinician judges that the subject is unsafe to enroll in the study or the subject cannot answer questions or follow instructions to fulfill the study

Any known cardiac or pulmonary disease

A woman with pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07-29; Primary Completion 2014-01-06 (Actual); Study Completion 2014-01-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are parameters representing gait performance such as maximum/self-selected walking speed, cadence, stride length, Time Up and Go test scores and Dynamic Gait Index scores.

SECONDARY OUTCOMES:
The secondary outcome measures are physical and cognitive effort exerted during the training. Physical effort will be measured by grip strength. Cognitive effort will be estimated by Letter Number Sequence test.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Campbell M, Parry A. Balance disorder and traumatic brain injury: preliminary findings of a multi-factorial observational study. Brain Inj. 2005 Dec;19(13):1095-104. doi: 10.1080/02699050500188898. PMID 16286323
- [Background] Katz-Leurer M, Rotem H, Lewitus H, Keren O, Meyer S. Relationship between balance abilities and gait characteristics in children with post-traumatic brain injury. Brain Inj. 2008 Feb;22(2):153-9. doi: 10.1080/02699050801895399. PMID 18240044
- [Background] Kerrigan DC, Bang MS, Burke DT. An algorithm to assess stiff-legged gait in traumatic brain injury. J Head Trauma Rehabil. 1999 Apr;14(2):136-45. doi: 10.1097/00001199-199904000-00004. PMID 10191372